CLINICAL TRIAL: NCT06194552
Title: A Multiple Ascending Dose, Phase 1, Double-Blind, Study to Investigate the Safety and Pharmacokinetics of NTRX-07 in Healthy Volunteers and Patients With Early Alzheimer's Disease (AD), With an Exploratory Fed-Fasted Assessment
Brief Title: A Multiple Dose Study of the Safety and Pharmacokinetics of NTRX-07
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroTherapia, Inc. (Industry)
Collaborators: CRU Early Phase Unit Kistarcsa (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTRX-C102
Record Dates: First submitted 2023-10-23; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer Disease
Keywords: CB2
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- NTRX-07 Low Dose Normal Volunteers (Experimental): NTRX-07 administered orally once per day for 7 days
  Interventions: Drug: NTRX-07
- NTRX-07 Mid Dose Normal Volunteers (Experimental): NTRX-07 administered orally once per day for 7 days
  Interventions: Drug: NTRX-07
- NTRX-07 High Dose Normal Volunteers (Experimental): NTRX-07 administered orally once per day for 7 days
  Interventions: Drug: NTRX-07
- NTRX-07 High Dose Alzheimer's Participants (Experimental): NTRX-07 administered orally once per day for 7 days
  Interventions: Drug: NTRX-07
- Placebo Control (Placebo Comparator): Placebo administered orally once per day for 7 days
  Interventions: Drug: Placebo
- Mid Dose Fed (Experimental): NTRX-07 administered orally once with high fat meal
  Interventions: Drug: NTRX-07

INTERVENTIONS:
Drug: NTRX-07 — Investigational orally administered CB2 agonist
  Other Names: MDA7
  Arms: Mid Dose Fed; NTRX-07 High Dose Alzheimer's Participants; NTRX-07 High Dose Normal Volunteers; NTRX-07 Low Dose Normal Volunteers; NTRX-07 Mid Dose Normal Volunteers
Drug: Placebo — Matched placebo administered orally
  Arms: Placebo Control

SUMMARY:
This is a Phase 1, Randomized, Placebo-Controlled, Modified Parallel Design Multiple Ascending Dose Study of NTRX 07 to Assess Safety and Tolerability and Pharmacokinetics in Adult Healthy Volunteers and Subjects with MCI or Early AD. In addition, an exploratory study of the effect of a high fat meal was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 45 80 years of age inclusive, at the time of signing the informed consent
* Cohorts A-C participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Cohort D - AD as characterized by the following clinical, cognitive, and functional criteria.

  * Diagnosis of a clinical syndrome of cognitive impairment consistent with prodromal AD per International Working Group (IWG) diagnostic criteria or mild AD per National Institute on Aging - Alzheimer's Association (NIAA-AA) diagnostic criteria
  * Self or informant report of memory decline
  * Mini-Mental State Examination (MMSE) scores between 18-27 inclusive within the last 4 months
  * Objective memory loss by education-adjusted Wechsler Memory Scale Logical Memory II consistent with mild cognitive impairment with Alzheimer's disease (MCI AD) or mild AD
  * Absence of significant levels of impairment in other cognitive assessments
* Cohort D - Previous brain imaging study, such as magnetic resonance imaging (MRI) and/or computed tomography (CT), consistent with a diagnosis of probably AD without any other clinically significant co-morbid pathologies within 12 months prior to the Screening Visit. If there has been a significant change in clinical status suggestive of stroke or other possible central neurological disease with onset between the time of the last MRI or CT and the Screening evaluation, the scan should be repeated during Screening procedures if considered appropriate by the Investigator OR Screening cerebrospinal fluid (CSF) results consistent with the presence of amyloid pathology.
* Cohort D - No active depression and a Geriatric Depression Score of <6.
* Cohort D - Absence of other (non-AD) types of dementia.
* Cohort D - Participants previously enrolled in an AD clinical trial involving a disease modifying or symptomatic therapeutic agent may enroll in this study if treatment with the symptomatic therapeutic agent ended more than 6 months before the first dose of NTRX 07-SDD in this study.
* Body weight within 55 110 kg and body mass index (BMI) within the range 18 35 kg/m2 (inclusive)
* Male or Female
* The effects of NTRX 07 on pregnancy, fetal development, and excretion in breast milk is currently unknown. Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the subject information sheet, informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Reported history or presence of clinically significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data. Participants with stable well controlled conditions may be accepted on review with the Investigator and sponsor.
* Reported current or chronic history of clinically significant liver disease. This includes but is not limited to hepatitis virus infections, drug- or alcohol-related liver disease, nonalcoholic steatohepatitis, autoimmune hepatitis, hemochromatosis, Wilson's disease, α-1 antitrypsin deficiency, primary biliary cholangitis, primary sclerosing cholangitis, or any other liver disease considered clinically significant by the investigator.
* Reported hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Cohort D - Reside in a nursing home or assisted care facility with need for direct continuous medical care and nursing supervision. Participant may reside in such facilities provided continuous direct medical care is not required.
* Cohort D - Unable to provide for self for basic activities of daily living.
* Cohort D - Major structural brain disease by reported history or chart review (eg, ischemic infarcts, subdural hematoma, hemorrhage, hydrocephalus, brain tumors, multiple subcortical ischemic lesions, or a single lesion in a critical region eg, thalamus, hippocampus).
* Any other reported history of central nervous system (CNS) trauma (eg, contusion), or infections that affect brain function (eg, human immunodeficiency virus [HIV], syphilis), history of seizures
* Diagnosis of schizophrenia
* Any reported history from patient, family, or on supplied chart review or current suicide risk
* Cohort D - Diagnosis of a dementia-related CNS disease other than AD (eg, Parkinson's Disease, Huntington's Disease, frontotemporal dementia, multi-infarct dementia, dementia with Lewy bodies, normal pressure hydrocephalus)
* Reported past or intended use of over-the-counter or prescription medication including herbal medications within 7 days prior to dosing. Specific medications listed in Section Concomittant Therapy may be allowed.
* Reported treatment with biologic agents (such as monoclonal antibodies including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing.
* Current enrollment or past participation within the last 30 days before signing of consent in any other clinical study involving an investigational study intervention or any other type of medical research.
* Alanine transaminase (ALT) or aspartate transaminase (AST) >1.5 x upper limit of normal (ULN)
* Total bilirubin >1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if total bilirubin is fractionated and direct bilirubin <35%)
* QTcF >450 msec for male participants or >470 msec for female participants
* Positive prestudy drug/alcohol screen
* Positive HIV antibody test
* Clinical laboratory findings outside the normal range and determined by the investigator or medical monitor to be clinically significant.
* Clinically significant abnormalities on screening EEG which may indicate an increased risk of seizure liability.
* Reported sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study
* Reported regular use of known drugs of abuse within the past 3 years.
* Presence of any contraindication to venous blood sampling for pharmacokinetic analyses.
* Positive SARS-CoV-2 test or hepatitis panel (including hepatitis B surface antigen [HBsAg] or hepatitis C virus antibody [anti-HCV]), or a positive HIV antibody screen
* Legal incapacity or limited legal capacity
* Participation in a clinical trial within 30 days prior to product administration.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events | From admission to discharge, up to 2 weeks
  AEs observed and recorded according to MEDRA

SECONDARY OUTCOMES:
Time to Maximum Concentration of NTRX-07 NTRX-07 | Day 1 and Day 7
  Pharmacokinetic profile of NTRX-07
Maximum Concentration of NTRX-07 NTRX-07 | Day 1 and Day 7
  Pharmacokinetic profile of NTRX-07
Area Under the Plasma Concentration Versus Time Curve (AUC) NTRX-07 | Day 1 and Day 7
  Pharmacokinetic profile of NTRX-07

OTHER OUTCOMES:
Plasma levels of neuro-inflammatory biomarkers | Day 1 and Day 7
  TNF-α, IL-1β, IL-6, IL-2, YKL-40, sTREM2, Aβ40, Aβ42, phospho-tau, Neurogranin, synaptotagmin-1, NfL - pg/ml
Plasma levels of high-sensitivity C-reactive protein (CRP) | Day 1 and Day 7
  high sensitivity CRP - ng/ml
MOCA Montreal Cognitive Assessment | Day 1 and Day 7
  Cognitive changes on patient-reported outcomes - Scored 0-30, higher is better
MMSE - Mini-Mental Status Exam | Day 1 and Day 7
  Cognitive changes on patient-reported outcomes - Scored 0-30, higher is better
ADAS-COG - Alzheimer's Disease Assessment Scale - Cognitive Scale | Day 1 and Day 7
  Cognitive changes on patient-reported outcomes - Scored 0-70, higher is worse

CONTACTS AND LOCATIONS:
Locations (2):
- NeuroTherapia, Gates Mills, Ohio, United States
- CRU Early Phase Unit Kistarcsa, Kistarcsa, Hungary

IPD SHARING:
Plan to Share IPD: No